CLINICAL TRIAL: NCT03943498
Title: Treatment of Established Chemotherapy-Induced Neuropathy With Fingolimod: A Pilot Trial
Brief Title: Fingolimod in Treating Patients With Chemotherapy-Induced Neuropathy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC18C2; NCI-2019-02742 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC18C2 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Numbness; Pain; Tingling
MeSH Terms: conditions — Hypesthesia; Pain; Paresthesia | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Fingolimod) (Experimental): Patients receive 0.5 mg dose of Fingolimod PO QD for 4 weeks.
  Take your Fingolimod approximately every 24 hours
  Interventions: Drug: Fingolimod; Drug: Fingolimod Hydrochloride; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Fingolimod — Given PO daily for 4 weeks
Drug: Fingolimod Hydrochloride — Given PO
  Other Names: FTY-720; FTY720; Gilenya
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial studies how well fingolimod works in treating patients with chemotherapy-induced nerve pain (neuropathy). Fingolimod acts by suppressing immune reactions in the brain. This study is being done to see if fingolimod can reduce neuropathy caused by chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether fingolimod markedly improves symptoms in patients with established (chemotherapy-induced peripheral neuropathy) CIPN.

II. To evaluate the tolerability of fingolimod in these treated patients.

OUTLINE:

Patients receive fingolimod orally (PO) once daily (QD) for 4 weeks.

After completion of study treatment, patients are followed up every month for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Pain or symptoms of CIPN of >= 3 months duration, for which the patient wants intervention.

  * NOTE: Neurotoxic chemotherapy must have been completed >= 6 months (186 days) prior to registration and there must be no further planned neurotoxic chemotherapy for > 6 months after registration.
* Tingling, numbness or pain was at least a four out of ten problem during the week prior to registration, on a 0-10 scale where zero was no problem and ten was the worst possible problem (patient verbal report to clinician).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2.
* Negative pregnancy test done =< 14 days prior to registration, for persons of childbearing potential only.
* Provided written informed consent.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Life expectancy >= 6 months.

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons.
  * Nursing persons.
  * Persons of childbearing potential who are unwilling to employ adequate contraception.
* Previous diagnosis of diabetic or other peripheral neuropathy.
* Current or previous use of fingolimod.
* History of the following preexisting conditions: ischemic heart disease, cardiac arrest, cerebrovascular disease, uncontrolled hypertension, symptomatic bradycardia, macular edema, recurrent syncope, severe untreated sleep apnea, herpes simplex virus (HSV) varicella zoster (VZV), chronic hepatitis, tuberculosis, fungal infections, skin cancer, or diabetes.
* Myocardial infarction, unstable angina, stroke, transient ischemic attack (TIA), decompensated heart failure requiring hospitalization or class III/IV heart failure =< 6 months prior to registration.
* History or presence of Mobitz type II second degree or third degree atrioventricular (AV) block or sick sinus syndrome, unless patient has a functioning pacemaker.
* History of hypersensitivity reaction to fingolimod or any of the excipients including rash, urticarial, and angioedema upon treatment initiation.
* Baseline corrected QT (QTc) interval >= 450 ms (on patient electrocardiography [EKG]).
* Concurrent use of a class Ia or III antiarrhythmic drug.
* Drugs with a known risk of torsades de pointes.
* Concurrent use of beta blockers, calcium channel blockers, or digoxin.
* Use of immunosuppressive or immune-modulating therapies that may have immunosuppressive effects.
* Immunocompromised patients including patients known to be human immunodeficiency virus (HIV) positive.
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection.
  * Unstable angina pectoris.
  * Cardiac arrhythmia.
  * Or psychiatric illness/social situations that would limit compliance with study requirements.
* Family history of genetic/familial neuropathy.
* Currently receiving another agent to treat CIPN, such as duloxetine, gabapentin or pregabalin, and not willing to be weaned off of these medications prior to therapy initiation.
* History of peripheral neuropathy prior to receiving neurotoxic chemotherapy.
* Received a vaccine (inactivated) =< 2 weeks prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Serially measured total sensory neuropathy scores | Baseline up to 3 months post treatment
  Will be obtained from the 6 individual Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20 (QLQ-CIPN20) questions that quantify numbness, tingling, and pain in the fingers (or hands) and toes (or feet). The hypothesis will be tested with the two-sided one-sample t-test at a significance level of 10% reduction. In the event that the distribution of the within-patients change from baseline in total sensory neuropathy scores is not approximately normally distributed, then variable transformation or a nonparametric one-sample Wilcoxon signed-rank test will be considered as alternative approaches.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) of fingolimod | Up to 4 weeks
  The constellation of AEs as scored using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0) will be summarized by reporting the number and percentage of patients. Specifically, to evaluate the AE profiles, the maximum grade for each type of AE are recorded for each patient and data listings and frequency tables are clinically reviewed to determine overall patterns, including AE attribution (possible, probable, and definite) to fingolimod. Sensory neuropathy will be graded as none, mild, moderate, and severe. The percentage of patients experiencing an improvement in sensory neuropathy from baseline using NCI CTCAE v5.0 will be calculated with the exact 90% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Loprinzi, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - The Ohio State University, Columbus, Ohio

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03943498/ICF_000.pdf